CLINICAL TRIAL: NCT02392429
Title: Early Assessment of Treatment Response in AML Using FLT PET/CT Imaging
Brief Title: FLT PET/CT in Measuring Response in Patients With Previously Untreated Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCI-2015-00328; NCI-2015-00328 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAI141; EAI141 (Other: ECOG-ACRIN Cancer Research Group); EAI141 (Other: CTEP); U10CA180820 (NIH); U10CA180827 (NIH)
Record Dates: First submitted 2015-03-18; First posted 2015-03-19 (Estimated); Results first posted 2024-08-06 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling; Biopsy; Drug Therapy; Cytarabine; alovudine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (anthracycline, cytarabine, FLT PET/CT) (Experimental): Patients receive anthracycline IV on days 1-3 and cytarabine IV on days 1-7 for up to 2 courses. Patients then undergo FLT PET/CT within 3 days before or after the nadir bone marrow biopsy (between days 10-17 after initiation of first induction cycle and prior to reinduction). Patients may undergo an optional FLT PET/CT prior to induction chemotherapy if it does not interfere with commencement of treatment. Patients also undergo bone marrow biopsy and aspiration and blood sample collection during screening and on the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Chemotherapy; Procedure: Computed Tomography; Drug: Cytarabine; Other: Fluorothymidine F-18; Other: Laboratory Biomarker Analysis; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Chemotherapy — Given anthracycline IV
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
Procedure: Computed Tomography — Undergo FLT PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Other: Fluorothymidine F-18 — Undergo FLT PET/CT
  Other Names: 18F-FLT; 3'-Deoxy-3'-(18F) Fluorothymidine; 3'-deoxy-3'-[18F]fluorothymidine; ALOVUDINE F-18; Fluorothymidine F 18
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Positron Emission Tomography — Undergo FLT PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase II trial studies fluorothymidine F 18 (FLT) positron emission tomography (PET)/computed tomography (CT) in measuring response in patients with previously untreated acute myeloid leukemia. FLT is a radioactive substance that may "light up" where cancer is in the body. FLT is injected into the blood and builds up in cells that are dividing, including cancer cells. Diagnostic procedures, such as PET/CT, may help measure a patient's response to earlier treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the negative predictive value (NPV) of post-treatment FLT PET/CT imaging for complete remission (CR) in patients receiving induction chemotherapy for acute myeloid leukemia (AML).

SECONDARY OBJECTIVES:

I. To evaluate the positive predictive value (PPV) of post-treatment FLT PET/CT imaging for complete remission.

II. To estimate the sensitivity and specificity of post-treatment FLT PET/CT imaging for detecting complete remission.

III. To correlate FLT PET/CT imaging with biologic correlates (minimal residual disease [MRD] assessment) IV. To correlate FLT PET/CT imaging with relapse-free survival and overall survival.

EXPLORATORY OBJECTIVES:

III. To evaluate pre-treatment FLT PET/CT imaging as a predictor of complete remission.

IV. To evaluate the change between pre-treatment and post-treatment FLT PET/CT imaging as a predictor of complete remission.

OUTLINE:

Patients receive anthracycline intravenously (IV) on days 1-3 and cytarabine IV on days 1-7 for up to 2 courses. Patients then undergo FLT PET/CT within 3 days before or after the nadir bone marrow biopsy (between days 10-17 after initiation of first induction cycle and prior to reinduction). Patients may undergo an optional FLT PET/CT prior to induction chemotherapy if it does not interfere with commencement of treatment. Patients also undergo bone marrow biopsy and aspiration and blood sample collection during screening and on the trial.

After completion of study, patients are followed up at day 28-35, and then up to 1 year beyond the end of study accrual period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients must have previously untreated AML and be candidates for intensive induction chemotherapy; patients are allowed to have had prior hydroxyurea
* Patients must not have acute promyelocytic leukemia (APL) and must not have evidence of t(15;17)(q22;q21)
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3 (restricted to ECOG performance status [PS] 0-2 if age > 70 years)
* Patients must have left ventricular ejection fraction (LVEF) > 45% or within institutional normal limits
* Patients must be able to lie still for a 1.5 hour PET scan
* Patient must NOT have a history of allergic reaction attributable to compounds of similar chemical or biologic composition to 18F-fluorothymidine
* Patient must NOT weigh more than the maximum weight limit for the PET/CT table for the scanner(s) to be used at each center
* The patient is participating in the trial at an institution which has agreed to perform the imaging research studies, completed the ECOG-American College of Radiology Imaging Network (ACRIN) defined scanner qualification procedures and received ECOG-ACRIN approval as outlined
* Women must not be pregnant or breast-feeding; all females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2016-04-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-02-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jeraj, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (11):
- United States (11):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on December 9, 2015 and finished accrual on October 16, 2018 after enrolling 87 participants from 9 institutions
Period: Screening
Arm/Group | Diagnostic (Anthracycline, Cytarabine, FLT PET/CT)
Started | 102
Completed | 87
Not Completed | 15
Not completed — Screen failure | 15
Period: Enrolled Participants
Arm/Group | Diagnostic (Anthracycline, Cytarabine, FLT PET/CT)
Started | 87
Optional Pre-treatment FLT PET/CT | 15
Completed | 71
Not Completed | 16
Not completed — Ineligible due to disease | 3
Not completed — Withdrawal by Subject | 4
Not completed — Post-treatment FLT PET/CT scan not completed | 9
Period: Evaluable
Arm/Group | Diagnostic (Anthracycline, Cytarabine, FLT PET/CT)
Started | 71
Completed | 61
Not Completed | 10
Not completed — Death | 5
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — remission bone marrow biopsy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Anthracycline, Cytarabine, FLT PET/CT)
Number analyzed (Participants) | 87
Age, Continuous [Mean (Full Range); unit: years] | 59 [21 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 80
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 77
  More than one race | 1
  Unknown or Not Reported | 4
Leukemia classification [Count of Participants; unit: Participants]
  AML with myelodysplasia-related changes | 25
  Other AML | 62

OUTCOME MEASURES:

1. Primary Outcome: Negative Predictive Value of Post-treatment Fluorothymidine F 18 (FLT) Positron Emission Tomography (PET)/Computed Tomography (CT) Imaging for Complete Remission (CR) in Comparison With Blast Counts From Bone Marrow Biopsy (BMBX)
Description: Three imaging parameters (standardized uptake value [SUV]mean, SUVmax, heterogeneity of FLT uptake [SUVhetero]) will be measured from an FLT PET/CT scan and SUVmax will be the primary endpoint. Higher values of SUVmax assume to indicate a non-response the therapy and a cut point of 7 (SUVmax >7) will be used as the threshold indicating a negative scan. The binomial proportion of negative predictive value (NPV) and the corresponding exact confidence intervals will be calculated. In addition, the calculated NPV will be tested against the null hypothesis to see if it's significantly larger than 0.64 (NPV of day-14 BMBX in CR prediction).
  CR:Complete remission CRi: Complete remission with incomplete platelet recovery LFS: Leukemia-free state Non-responders defined as Not (CR,CRi,or LFS)
  Negative predictive value (NPV) of the post-treatment FLT PET/CT scan is Probability ((not CR,CRi,or LFS) │ SUVmax >7 )
Time Frame: Up to day 35
Measure: Number (95% Confidence Interval); unit: Proportion of Negative scans
Groups:
- Diagnostic (Anthracycline, Cytarabine, FLT PET/CT) Negative: Patients with a Negative FLT PET (High FLT uptake defined as SUVmax > 7)
Arm/Group | Diagnostic (Anthracycline, Cytarabine, FLT PET/CT) Negative
Number analyzed (Participants) | 15
Proportion of Negative scans | 0.20 [0.04 to 0.48]
Statistical Analysis 1: Comparison: Diagnostic (Anthracycline, Cytarabine, FLT PET/CT) Negative; Test type: Non-Inferiority — we tested the null hypothesis that the NPV of the post-treatment FLT PET/CT scan was less than or equal to the NPV of the day 14 nadir bone marrow biopsy (estimated to be 0.64 by Hussein et al) against the one-sided alternative hypothesis that the NPV was greater than 0.64 using the exact binomial test; p > 0.99, binomial exact test

2. Secondary Outcome: Positive Predictive Value (PPV) of Post-treatment FLT PET/CT Imaging for Complete Remission
Description: The binomial proportion of PPV and the corresponding exact confidence intervals will be calculated. In addition, the calculated PPV will be tested to see if it's significantly larger than 0.79 (PPV of day-14 BMBX in CR prediction).
Time Frame: Up to day 35
Measure: Number (95% Confidence Interval); unit: Proportion of Positive Scans
Groups:
- Diagnostic (Anthracycline, Cytarabine, FLT PET/CT) Positive: Patients with a Positive FLT PET (Positive FLT uptake defined as SUVmax <= 7)
Arm/Group | Diagnostic (Anthracycline, Cytarabine, FLT PET/CT) Positive
Number analyzed (Participants) | 46
Proportion of Positive Scans | 0.89 [0.76 to 0.96]
Statistical Analysis 1: Comparison: Diagnostic (Anthracycline, Cytarabine, FLT PET/CT) Positive; Test type: Non-Inferiority — we tested the null hypothesis that the PPV of the post-treatment FLT PET/CT scan was less than or equal to the PPV of the day 14 nadir bone marrow biopsy (estimated to be 0.79by Hussein et al) against the one-sided alternative hypothesis that the PPV was greater than 0.79 using the exact binomial test; p = 0.06, binomial exact test

3. Secondary Outcome: Sensitivity of Post-treatment FLT PET/CT for Detecting Complete Remission (a Clinical Response of CR, CRi, or LFS )
Description: The binomial proportions and the corresponding exact confidence intervals will be calculated for sensitivity estimation where
  FLT Test :
  Negative: SUV >7; Positive: SUV<=7
  Clinical Response:
  Negative: not (CR, CRi, or LFS); Positive (Responders): CR, CRi, or LFS
Time Frame: Up to day 35
Population: Responders: Patients with a Positive clinical response: CR, CRi, or LFS.
Measure: Number (95% Confidence Interval); unit: Proportion of Responders
Arm/Group | Diagnostic (Anthracycline, Cytarabine, FLT PET/CT)
Number analyzed (Participants) | 53
Proportion of Responders | 0.77 [0.64 to 0.88]

4. Secondary Outcome: Specificity of Post-treatment FLT PET/CT for Detecting Complete Remission
Description: The binomial proportions and the corresponding exact confidence intervals will be calculated for specificity estimation.
  Test response:
  Negative: SUV >7; Positive: SUV<=7
  Clinical Response = Complete remissions:
  Negative (Non-Responders): not (CR, CRi, or LFS); Positive (Responders): CR, CRi, or LFS
Time Frame: Up to day 35
Population: Non-Responders: No Clinical Response for any of CR, CRi, or LFS.
Measure: Number (95% Confidence Interval); unit: Proportion of Non-Responders
Arm/Group | Diagnostic (Anthracycline, Cytarabine, FLT PET/CT)
Number analyzed (Participants) | 8
Proportion of Non-Responders | 0.38 [0.09 to 0.76]

5. Secondary Outcome: FLT PET/CT Imaging Parameters With Biologic Correlates (Minimal Residual Disease Assessment)
Description: FLT PET/CT imaging features will be compared with biologic correlates (minimal residual disease [MRD] assessment).
Time Frame: Up to day 35
Reporting Status: Not Posted

6. Secondary Outcome: FLT PET/CT Imaging to Predict Relapse-free Survival
Description: compare the Recurrence-Free Survival (RFS) between positive and negative post-treatment FLT PET/CT scans, where an SUVmax less than or equal to 7 (i.e., low FLT uptake) was considered a positive result, and an SUVmax greater than 7 (i.e., high FLT uptake) was a negative result.
  Participants were followed for survival outcomes until study closure when the last participant has been followed for 1 year after study enrollment.
  The relapse endpoint included both reappearance of blasts in the blood; and presence of more than 5% blasts not attributable to another cause Time-to-relapse was measured from the date of the remission bone marrow biopsy to the date of first recurrence or death, whichever came first.
  RFS was only evaluable for participants with a clinical response of CR, CRi, or LFS at the remission bone marrow biopsy.
Time Frame: Up to day 35 and up to 4 years for RFS
Population: Only participants with a clinical response of CR, CRi, or LFS at the remission bone marrow biopsy (ie., where RFS is evaluable)
Measure: Count of Participants; unit: Participants
Groups:
- FLT PET/CT Positive: Patients with a Positive FLT PET (Positive FLT uptake defined as SUVmax <= 7)
- FLT PET/CT Negative: Patients with a Negative FLT PET (Negative FLT uptake defined as SUVmax >7)
Arm/Group | FLT PET/CT Positive | FLT PET/CT Negative
Number analyzed (Participants) | 41 | 12
Participants
  Recurrence | 25 | 6
  Disease-free | 16 | 6
Statistical Analysis 1: Comparison: FLT PET/CT Positive vs FLT PET/CT Negative; Kaplan-Meier curves were constructed for the positive and negative scan groups, and the null hypothesis that the survival distributions of the two groups were equal was tested using the log-rank test; Test type: Equivalence — no margin was assumed; p = 0.68, log-rank test

7. Secondary Outcome: FLT PET/CT Imaging to Predict Overall Survival
Description: compare the Overall Survival (OS) between positive and negative post-treatment FLT PET/CT scans, where an SUVmax<= 7 (i.e., low FLT uptake) was considered a positive result, and an SUVmax > 7 (i.e., high FLT uptake) was a negative result.
  Participants were followed for survival outcomes until study closure when the last participant has been followed for 1 year after study enrollment.
Time Frame: Up to day 35 and up to 4 years for RFS
Population: All participants who received an FLT PET/CT scan were included in the OS analysis,
Measure: Count of Participants; unit: Participants
Arm/Group | FLT PET/CT Positive | FLT PET/CT Negative
Number analyzed (Participants) | 51 | 20
Participants
  Survivors | 37 | 10
  Non-survivors | 14 | 10
Statistical Analysis 1: Comparison: FLT PET/CT Positive vs FLT PET/CT Negative; [analysis description as in outcome 6, analysis 1]; Test type: Equivalence — no margin was assumed; p = 0.08, log-rank test

ADVERSE EVENTS:
Time Frame: 5 years
Description: Within 24 hours after administration of FLT, all serious AEs worsening or emergent after FLT administration were considered reportable.
  After 24 hours after administration of FLT, all serious AEs that were attributed as possibly, probably, or definitely related to the study procedure were considered reportable.
Arm/Group | Diagnostic (Anthracycline, Cytarabine, FLT PET/CT)
All-Cause Mortality (participants affected / at risk) | 30/87
Serious Adverse Events (participants affected / at risk) | 24/87
Other Adverse Events (participants affected / at risk) | 4/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (Anthracycline, Cytarabine, FLT PET/CT) (N=87)
Abdominal pain (Gastrointestinal disorders) | 1 (1) — 10000081: Gastrointestinal disorders
Allergic reaction (Immune system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Death NOS (General disorders) | 7 (7)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Multi-organ failure (General disorders) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Progressive AML disease (Blood and lymphatic system disorders) | 1 (1)
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Troponin elevated (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (Anthracycline, Cytarabine, FLT PET/CT) (N=87)
Fever (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT02392429/Prot_SAP_000.pdf